CLINICAL TRIAL: NCT06459713
Title: The Use of Multiplex Respiratory Polymerase Chain Reaction Test in Patient With Diabetes Mellitus Who Have a Newly Diagnosed of Community-acquired Pneumonia
Brief Title: Multiplex Respiratory PCR Results in Diabetic Pneumonia Cases
Acronym: PCR
Status: Completed | Type: Observational
Sponsor: Hisar Intercontinental Hospital (Other)
Responsible Party: Principal Investigator, Bekir Sami Uyanık, Clinical Biochemistry, Hisar Intercontinental Hospital
Other Study IDs: HisarOD
Record Dates: First submitted 2024-05-31; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-05

CONDITIONS: Multiplex Respiratory PCR Results in Diabetic Pneumonia Cases
Keywords: pneumonia, multiplex respiratory PCR test
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — nasopharyngeal swab samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiplex respiratory PCR test results of the groups: This single center retrospective observational study was conducted in Hisar Hospital Intercontinental between September 2021 and June 2023
  Interventions: Diagnostic Test: multiplex respiratory polymerase chain reaction test
- we evaluated the importance of respiratory PCR in CAP: Subjects who had an infection other than pneumonia, and had a diagnosis of malignancy, transferred to intensive care unit and pregnant women were excluded.
  Interventions: Diagnostic Test: multiplex respiratory polymerase chain reaction test

INTERVENTIONS:
Diagnostic Test: multiplex respiratory polymerase chain reaction test — According to our hospital policy, nasopharyngeal swab samples are collected by the clinicians and transported to the Clinical Microbiology Laboratory of the hospital in 10 minutes. The samples are analyzed in 2 hours and the samples were measured by Thermo Fisher / Applied Biosystems Quant Studio-5 for reverse transcription-polymerase chain reaction (RT-PCR) testing to detect multiplex respiratory agents

SUMMARY:
Multiplex respiratory polymerase chain reaction (PCR) test has gained wide acceptance as an alternative to conventional culture methods for the detection of the causative agent of community-acquired pneumonia (CAP). The aim of this study is to evaluate the positivity and to determine the causative agent of CAP using multiplex respiratory PCR test in patients with diabetes mellitus.

DETAILED DESCRIPTION:
A total of 151 adults diagnosed with CAP were enrolled. Group 1 composed of patients who had diabetes (n=42) and group 2 consisted of patients who did not have diabetes (n=109). Demographic and clinical data of the subjects were collected and compared statistically.

The multiplex respiratory PCR test positivity of group 1 was statistically higher than group 2 (p=0.004). The most identified nasopharyngeal pathogen was SARSCoV2 in group 1, whereas in group 2, the most prevalent agent was Streptococcus pneumoniae (p=0.002, p=0.628). Furthermore, the amount of procalcitonin, CRP, neutrophil counts and the ratio of neutrophil-to-lymphocyte ratio (NLR) and CRP-to-lymphocyte (CLR) ratio on admission were statistically higher in group 1 than groups 2 (p=0.012, p=0.002, p<<0.001, p=0.001, p=0.001).

Diabetic patients are at greater risk for developing CAP. Therefore, early detection and prompt treatment is crucial for diabetic patients with CAP to avoid morbidity and mortality. Multiplex respiratory PCR test is an important method for identifying the causative agent of CAP rapidly.

ELIGIBILITY:
Inclusion Criteria:

In this study, a population of 190 people over the age of 18 were searched in terms of suitability for this work , who diagnosed with CAP after admission to the Department of Chest Diseases by using a multiplex respiratory PCR test.

Exclusion Criteria:

Subjects who had an infection other than pneumonia, and had a diagnosis of malignancy, transferred to intensive care unit and pregnant women were excluded.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: After the exclusion criteria applied, remaining 151 patients were enrolled in the study. Of the 151 subjects, 42 (27.8%) who were followed up with the confirmed diagnosis of type 2 diabetes mellitus constituted group 1 and 109 (72.2%) ones who did not have a diagnosis of type 2 diabetes mellitus named as group 2. -
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Diabetic patients are at greater risk for developing CAP. Multiplex respiratory PCR test is an important method for identifying the causative agent of CAP rapidly. | September 2021 and June 2023

CONTACTS AND LOCATIONS:
Overall Officials: Yakup Tomak, Study Director — Hisar Intercontinental Hospital
Locations (1):
- Hisar Intercontinental Hospital, Istanbul, Turkey (Türkiye)